CLINICAL TRIAL: NCT01009502
Title: SHP2 as a Therapeutic Target For Myelodysplastic Syndrome: Phase I/II Trial of Sodium Stibogluconate in Myelodysplastic Syndrome
Brief Title: Phase I/II Trial of Sodium Stibogluconate in Myelodysplastic Syndrome
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding, never moved into the phase II portion that was originally planned.
Sponsor: Northwestern University (Other)
Collaborators: Robert H. Lurie Cancer Center (Other)
Responsible Party: Principal Investigator, Elizabeth Eklund, Elizabeth Eklund, MD, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 08H4; 2008-0807 (Other: University of Illinois at Chicago IRB); STU00005048 (Other: Northwestern University IRB); NCI-2010-02059 (Other: NCI CTRP#)
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Antimony Sodium Gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sodium stibogluconate (Experimental): Sodium stibogluconate 900 mg/m2/day will be given on Monday through Friday every other week for the first 16 weeks of the study (on the 1st, 3rd, 5th, 7th, 9th, 11th, 13th and 15th weeks). On the alternate weeks patients will not receive any study treatment.
  Interventions: Drug: sodium stibogluconate

INTERVENTIONS:
Drug: sodium stibogluconate — Sodium stibogluconate 900 mg/m2/day will be given on Monday through Friday every other week for the first 16 weeks of the study (on the 1st, 3rd, 5th, 7th, 9th, 11th, 13th and 15th weeks). On the alternate weeks patients will not receive any study treatment.

SUMMARY:
Sodium stibogluconate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

This was originally designed as a phase I/II trial studying the side effects of sodium stibogluconate and how well it works in treating patients with myelodysplastic syndromes. Unfortunately, due to funding issues, the phase II portion was never conducted.

DETAILED DESCRIPTION:
Patients receive sodium stibogluconate IV over 30 minutes on days 1-5 and 15-19. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients who respond to treatment may continue therapy until disease progression.

Patients undergo bone marrow aspiration, biopsy, and peripheral blood sample collection periodically for correlative laboratory studies.

After completion of study treatment, patients are followed up at 8 weeks.

The phase II portion of this trial was never conducted due to lack of funding.

ELIGIBILITY:
Inclusion Criteria:

* Documented myelodysplastic syndromes (MDS), including therapy-related MDS
* Meets 1 of the following criteria:

  * Refractory to prior azacitidine or decitabine
  * Did not tolerate treatment with azacitidine or decitabine due to cytopenias or other side effects
  * Not a candidate for azacitidine or decitabine due to cytopenias or other medical conditions that would contraindicate nucleoside analogues
  * Refused treatment with azacitidine or decitabine
* Life expectancy ≥ 16 weeks
* Not pregnant or nursing
* No B12 deficiency, folate deficiency, or pyridoxine responsive anemia as confirmed by relevant laboratory testing
* No prolongation of QTc or ventricular ectopic beats on EKG
* No evidence of cardiac disease
* No active infection AND afebrile
* More than 21 days since prior azacitidine or decitabine
* More than 21 days since other prior treatment for MDS (e.g., thalidomide, valproic acid, or other agents as part of a clinical trial)
* Prior cytokines (e.g., erythropoietin, G-CSF, and GM-CSF) allowed
* Prior chemotherapy and/or radiotherapy for solid tumors or lymphoma allowed provided there is no evidence of active disease from the prior malignancy

Exclusion Criteria:

* Prior treatment for leukemia (e.g., acute myeloid leukemia, chronic myelogenous leukemia, acute lymphocytic leukemia, or chronic lymphocytic leukemia)
* Concurrent cytokines
* Concurrent antileukemic treatment, including bone marrow transplantation and radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-07; Primary Completion 2012-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
determine the effect of SSG treatment on clinical parameters of MDS | Weeks 2 and 4 of each cycle for 24 Weeks then every other month for 6 months then every 3 months for 12 months then every 6 months for 2 years
  To determine the effect of SSG treatment on clinical parameters of MDS. This will include determination of cytopenias, bone marrow dysplasia, % myeloid blasts, transfusion frequency, incidence of infection and phagocyte function in MDS subjects pre and during treatment. Serum Sb levels will also be determined as an early indication of toxicity.
Determine the effect of SSG treatment on hematopoiesis in MDS subjects | Weeks 2 and 4 of each cycle for 24 Weeks then every other month for 6 months then every 3 months for 12 months then every 6 months for 2 years
  To determine the effect of SSG treatment on hematopoiesis in MDS subjects. This will include determination of cytokine hypersensitivity, apoptosis resistance, and altered expression of key HoxA10 and ICSBP target genes in the bone marrow of subjects pre and during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Eklund, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Jesse Brown VHA Medical Center, Chicago, Illinois